CLINICAL TRIAL: NCT06261944
Title: A Pivotal Multi-centre, Open-label, Two-part Clinical Investigation Confirming the Safety and Accuracy of the Glyconics-DS in Assessment of Glycated Nail Keratin in Individuals With Unknown Diabetes Status and Performance Evaluation of the Glyconics SW Package Delivering the Dichotomised Results
Brief Title: A Pivotal Clinical Investigation Confirming the Safety and Accuracy of the Glyconics-DS in Assessment of Glycated Nail Keratin in Individuals With Unknown Diabetes Status and Performance Evaluation of the Glyconics SW Package
Acronym: ANODE03
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glyconics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NIRDM-SXCIP03
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Pre-diabetes; Undiagnosed Diseases
MeSH Terms: conditions — Glucose Intolerance; Undiagnosed Diseases | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Intervention Model Description: Mass-screening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): All individuals will be screened for their diabetes risk / status (if previously undiagnosed)
  Interventions: Device: Near-infrared (NIR)

INTERVENTIONS:
Device: Near-infrared (NIR) — Near-infrared assessment of glycated keratin in middle fingernail

SUMMARY:
The main clinical study objective is to confirm the accuracy of the Glyconics-DS spectrometer when used in its intended medical purpose population, i.e., in individuals with unknown diabetes risk. Additionally, this investigation will serve as a pivotal performance evaluation for the associated software for correct delivery of the algorithm-based analysis of the individual diabetes risk. The study will be considered positive if the backend delivery of the chemometrics output is performed correctly as per the cloud-based analysis and its delivery represents the essential medical software to be evaluated in this investigation. The 'true' diabetes risk will be contrasted against values of an internal biomarker indicative of glycaemia, HbA1c, as measured based on standardised, certified methodology.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy adults (≥18 years of age) with unknown diabetes status willing to participate in and provide a written consent for the study
* Willingness to undertake assisted assessment of glycaemia: by both the NIR spectral measurements in a chosen middle fingernail, and HbA1c (blood sample)
* Individuals with at least one visually assessed undamaged, intact (preferably middle) fingernail.

Exclusion Criteria:

* Individuals with any known medical conditions impacting either of the assessment methodology for glycaemia, such as:

  * Severe forms of anaemia (diagnosed iron deficiency, sickle cell anaemia or similar).
  * Haemoglobinopathies or atypical haemoglobin subtypes not detectable by regular (local) laboratory assays for HbA1c.
  * Severe renal impairment (CKD stage III-IV) or decompensated hepatic disease.
  * Severe Vitamin D deficiency (diagnosed or measured 25(OH)D3 < 25 nmol/ml).
  * Known severe immunodeficiency such as HIV, malignancy or other chronic condition significantly impacting assessment of glycaemia.
  * Eating disorders (as per clinical assessment)
  * Recent (within 28 days) blood donation
  * Any other type of known diabetes than T2DM, if diagnosed (T1DM, GDM, MODY, etc.)
* Any structural, deviating and visually detectable deviations in the appearance of the (only/ to be assessed) middle fingernail potentially impacting the spectra measurement, including:

  * nail dystrophy or deformity
  * severe nail infections (onychomycosis causing visual changes in the appearance of the nail).
  * rare hereditable conditions impacting the structure of keratin.
  * mechanical damage or marks on the surface of the nail after removal of nail polish.
  * use of acrylic or gel nail decoration and polish, which cannot be removed with acetone (use of acetone necessitates a 15 min post-removal wash-out time)
* Any systemic or topical medication known to modify either the surface or structure of the nail or accuracy of HbA1c value.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-08-08 (Estimated)

PRIMARY OUTCOMES:
Dichotomised diabetes risk status | 10 seconds
  YELLOW: HbA1c value < 48 mmol/mol OR ORANGE: HbA1c value >= 48 mmol/mol.

SECONDARY OUTCOMES:
Sensitivity and specificity | 10 seconds
  HbA1c cut-off value of 48 mmol/mol (6.5%) and HbA1c cut-off value of 42 mmol/mol (6.0%)

CONTACTS AND LOCATIONS:
Overall Officials: Didac Mauricio, MD, PhD, Principal Investigator — Sant Pau Hospital
Locations (1):
- Sant Pau Hospital, Barcelona, Spain